CLINICAL TRIAL: NCT04594980
Title: An Open-Label Randomized Controlled Study of the Efficacy of Surgical Treatment in Patients With Single Level Lumbar Spinal Stenosis Using Minimally Invasive Decompression and Fusion and Traditional Open
Brief Title: Minimally Invasive Decompression and Fusion Versus Open for Degenerative Lumbar Stenosis
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: N.N. Priorov National Medical Research Center of Traumatology and Orthopedics (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: NS02-01
Record Dates: First submitted 2020-10-10; First posted 2020-10-20 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Lumbar Spinal Stenosis; Intervertebral Disc Degeneration
MeSH Terms: conditions — Spinal Stenosis; Intervertebral Disc Degeneration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Minimally invasive TLIF (Other): Patients will undergo a single level decompression and fusion using a minimally invasive technique. Followed posterior screw fixation is mandatory.
  Interventions: Procedure: lumbar fusion
- Open TLIF (Other): Patients will undergo a single level decompression and fusion using an open traditional technique. Followed posterior screw fixation is mandatory.
  Interventions: Procedure: lumbar fusion

INTERVENTIONS:
Procedure: lumbar fusion — Transforaminal Lumbar Interbody Fusion will be performed using minimally invasive approach or traditional open technique.

SUMMARY:
The purpose of this study is to determine the effectiveness of minimally invasive decompression and fusion over the traditional open decompression and fusion in patients with single-level lumbar stenosis caused by degenerative spondylolisthesis. Postoperative follow-up will continue for 12 months. Сlinical, safety, radiological and cost-effectiveness endpoints will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Age 40-75 years;
2. Neurogenic claudication or bilateral radiculopathy caused by single level combination of degenerative stenosis and spondylolisthesis confirmed by MRI at one level L3-L4 or L4-L5 or L5-S1;
3. Symptoms persisting for at least three months prior to surgery;
4. Given written Informed Consent Form;
5. Able and agree to fully comply with the clinical protocol and willing to adhere to follow-up schedule and requirements;
6. Oswestry Disability Index score of at least 40/100 at baseline;

Exclusion Criteria:

1. Bilateral foraminal stenosis requiring surgical decompression on both sides;
2. Degenerative spondylolisthesis Type 2B, 3 subtypes by Gille;
3. More than one symptomatic level requiring multi-level surgical decompression and/or fusion;
4. Any condition that cannot be treated with mini-invasive unilateral decompression and fusion;
5. Any contraindication or inability to undergo baseline and/or follow up MRI or X-ray as required per protocol;
6. Spondylolisthesis grade II or higher of any etiology;
7. Prior lumbar spinal fusion at any level;
8. Other non-degenerative spinal conditions that may have an impact on subject safety, wellbeing or the intent and conduct of the study;
9. History or presence of any other major neurological disease or condition that may interfere with the study assessments;
10. Severe arterial insufficiency of the legs or other peripheral vascular disease;
11. Previous enrollment in this study, current enrollment or plans to be enrolled in another study (in parallel to this study).

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2022-01-20 (Actual); Primary Completion 2024-02-27 (Actual); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Oswestry Disability Index (ODI) | 3 months
  To observe the change of ODI as compared to baseline through follow-up terms. min - 0, - the best result, patient is active; max - 50 - the worst result, patient is not physically active

SECONDARY OUTCOMES:
Change from baseline in Oswestry Disability Index (ODI) | Through 2 years
  To observe the change of ODI as compared to baseline through follow-up terms. min - 0, - the best result, patient is active; max - 50 - the worst result, patient is not physically active
Change from baseline in Numeric Pain Rating Score (NPRS) | Through 2 years
  To observe the change of NPRS as compared to baseline through follow-up terms (0 - no pain, 10 - unbearable pain)
Change from baseline in EuroQol Five-Dimensional descriptive system questionnaire (EQ-5D). | Through 2 years
  To observe the change of EQ-5D as compared to baseline through follow-up terms. It assesses 5 components related to aspects of life: mobility, self-care, activity in daily life, pain, anxiety or depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems.
Change from baseline in Douleur Neuropathique 4 (DN4) | Through 2 years
  To observe the change of DN4 as compared to baseline through follow-up terms. The scale result ranges 0-10 points. The sum > 4 points indicates the neuropathic component of pain
Change from baseline in The Health Transition Item from SF-36 (HTI Item) | Through 2 years
  To observe the change of HTI Item through follow-up terms. Patient's answers range from ''Much Better,'' ''Somewhat Better,'' ''About the Same,'' ''Somewhat Worse,'' to ''Much Worse.''
Change from baseline in Clinical Global Impression Of Change (CGIC) scale | Through 2 years
  To observe the change of CGIC through follow-up terms. The answers range from "-2 Significantly worse compared to Baseline" to "+2 Significantly improved compared to Baseline". 7-points scale indicates the patient's condition assessed by physician.
Cost-effectiveness | 14th day of hospital stay
  Total cost of surgical procedure (implanted system, the salary for surgery team) and the cost of patient's staying at the clinic before discharge.
Fusion rate success | 12 months and 24 months post op
  Interbody fusion rate on CT based on Tan grades
Surgery duration | Day of surgery
  Surgery duration, min
Reoperations rate | Through 2 years
  Incidence of reoperations
Pelvic Incidence | Through 2 years
  To observe the sagittal balance parameter - Pelvic Incidence - by sagittal scans of spine by X-Ray, in degrees
Change from baseline in Pelvic Tilt | Through 2 years
  To observe the sagittal balance parameter - Pelvic Tilt - by sagittal scans of spine by X-Ray compared to baseline, in degrees
Change from baseline in Global Lordosis Angle | Through 2 years
  To observe the sagittal balance parameter - Global Lordosis Angle - by sagittal scans of spine by X-Ray compared to baseline, in degrees
Change from baseline in Segmental Lordosis | Through 2 years
  To observe the sagittal balance parameter - Segmental Lordosis (the angle of treated level) - by sagittal scans of spine by X-Ray compared to baseline, in degrees
Change from baseline in Sagittal Vertical Axis | Through 2 years
  To observe the sagittal balance parameter - Sagittal Vertical Axis - by sagittal scans of spine by X-Ray compared to baseline, in mm
Adverse Events | Through 2 years
  Document Adverse Events (incl. adverse events related to device) occurrence throughout the study

CONTACTS AND LOCATIONS:
Locations (1):
- Priorov National Medical Research Center of Traumatology and Orthopedics, Moscow, Russia

IPD SHARING:
Plan to Share IPD: Yes
Data are available upon reasonable request. Please contact the corresponding author for detail.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: During the study conducting and during 5 years after
Access Criteria: The approval of institutional review board will be necessary

REFERENCES:
- [Derived] Leonova ON, Cherepanov EA, Krutko AV. MIS-TLIF versus O-TLIF for single-level degenerative stenosis: study protocol for randomised controlled trial. BMJ Open. 2021 Mar 5;11(3):e041134. doi: 10.1136/bmjopen-2020-041134. PMID 33674366